CLINICAL TRIAL: NCT02503852
Title: Subcutaneous Transplantation of Autologous Cell Enriched Adipose Tissue For Follicular Niche Stimulation in Early Stage Alopecia Androgenetica (STYLE): a Randomized, Blinded, Controlled Trial
Brief Title: STYLE -- A Trial of Cell Enriched Adipose For Androgenetic Alopecia
Acronym: STYLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerastem Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003-A-II
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-08

CONDITIONS: Alopecia, Androgenetic
Keywords: Female Pattern Baldness; Male Pattern Baldness; Genetic Alopecia; Androgenic Alopecia; Hair Loss
MeSH Terms: conditions — Alopecia | interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: Subjects arm randomized prior to liposuction 2:2:2:1 ratio to one of 4 Arms. Low Dose ADR, High Dose ADRC, non enriched fat only, and no fat (control normal saline).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization via manual treatment assignment by the unblinded Clinical Supply Manager prior to the start of liposuction.
  Subjects randomized into the study are assigned their study Arm corresponding to the next available number in the computer-generated randomization schedule. Dose preparation ios performed by designated unblinded qualified personnel and supplied to the blinded treating team.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fat + High Dose ADRC (Experimental): Kerastem Therapy includes micro-liposuction followed by subcutaneous scalp injection of purified adipose prepared with the Puregraft System + 1,000,000 ADRC prepared with the Celution System per square centimeter of scalp.
  Interventions: Device: Puregraft System; Device: Celution System; Procedure: Kerastem Therapy; Procedure: Liposuction
- Fat + Low Dose ADRC (Experimental): Kerastem Therapy includes micro-liposuction followed by subcutaneous scalp injection of purified adipose prepared with the Puregraft System + 500,000 ADRC prepared with the Celution System per square centimeter of scalp.
  Interventions: Device: Puregraft System; Device: Celution System; Procedure: Kerastem Therapy; Procedure: Liposuction
- Fat Alone (Active Comparator): Micro-liposuction followed by subcutaneous scalp injection of purified adipose prepared with the Puregraft System per square centimeter of scalp.
  Interventions: Device: Puregraft System; Procedure: Liposuction
- No Fat Control (Placebo Comparator): Micro-liposuction followed by subcutaneous scalp injection of normal saline per square centimeter of scalp.
  Interventions: Procedure: Liposuction

INTERVENTIONS:
Device: Puregraft System — The Puregraft System prepares purified adipose tissue for subcutaneous scalp injection.
  Arms: Fat + High Dose ADRC; Fat + Low Dose ADRC; Fat Alone
Device: Celution System — The Celution System prepares adipose derived regenerative cells (ADRCs) for subcutaneous scalp injection.
  Arms: Fat + High Dose ADRC; Fat + Low Dose ADRC
Procedure: Kerastem Therapy — The Kerastem Therapy is the subcutaneous scalp injection of purified adipose prepared with the Puregraft System enriched with ADRCs prepared from the Celution System.
  Arms: Fat + High Dose ADRC; Fat + Low Dose ADRC
Procedure: Liposuction — Tissue collection involving the micro-harvest of subcutaneous adipose tissue.

SUMMARY:
The primary objective of this study is to evaluate the safety and feasibility of the Celution and Puregraft Systems in the processing and preparation of an autologous fat graft enriched with adipose-derived regenerative cells (ADRCs) in the treatment of early alopecia androgenetica.

DETAILED DESCRIPTION:
The STYLE Trial is a prospective, randomized, multi-center device trial intended to evaluate the safety and efficacy of the Celution and Puregraft Systems in the processing and preparation of an autologous fat graft enriched with adipose-derived regenerative cells (ADRCs) in the treatment of early alopecia androgenetica. Patients may be included if they are undergoing an elective cosmetic liposuction. Following informed consent and screening evaluations, eligible subjects will undergo pre-operative testing. Subjects will then undergo a fat harvest using local anesthesia with or without conscious sedating. Subjects will be randomly assigned to receive a fat graft cell enriched with ADRCs (available in two different doses),a fat graft without cell enrichment using a visually-matched blood saline solution (fat alone control), or a saline injection (no-fat control) in a 2:2:2:1 ratio.

While undergoing liposuction, lipoaspirate will be processed in the Puregraft System to remove the lipoaspirate of impurities and in the Celution System to isolate and concentrate ADRCs. After the liposuction is completed), patients will have, under a ring block local anesthesia (see further description below), a subcutaneous scalp injection of either Puregraft purified autologous fat or saline (no-fat control) followed by a separate second injection, of either ADRCs (available in two different doses),a visually-matched blood saline solution (fat alone control), or saline (no-fat control) in a 2:2:2:1 ratio.

The STYLE Clinical Trial will have a sample size of 70 patients at up to eight (8) centers.

ELIGIBILITY:
Inclusion Criteria:

1. Males with a diagnosis of Alopecia Androgenetica
2. Females with a diagnosis of Alopecia Androgenetica
3. Males with hair loss consistent with Grades III, IIIA, III-Vertex, IV, IV-A, based on Norwood-Hamilton Scale (Figure 1)
4. Females with hair loss consistent with Grades I-3, I-4, II-1, II-2 based on the Savin Scale (Figure 2)
5. Provide written informed consent and comply with the study requirements
6. For women of childbearing potential: Negative pregnancy test at screening visit plus subject agrees to maintain two forms of contraception for the duration of the study.
7. Subject is willing to maintain a consistent hair length and natural hair color, without the use of any coloring agents, during the study period.
8. Ability to complete study procedures, patient surveys, and pictures.
9. Subject is ≥ 18 years of age.
10. Body Mass Index < 40kg/m2

Exclusion Criteria:

1. Subjects who have used minoxidil, or any oral or topical medication including over the counter and herbal medications for the treatment of hair loss within 6 months of study screening, or finasteride or dutasteride within 12 months of study screening
2. Treatment with an investigational product or procedure within 30 days or plans to participate in another clinical study
3. Subject who has previously failed or has been deemed non-responsive to a previous experimental hair loss treatment.
4. Subject must have no previous hair transplant, cell treatment, micro needling, or any other treatment in the last 6 months in the scalp.
5. Subject is currently suffering from an active autoimmune disease such as serum lupus erythematosus, or alopecia areata. Subject is currently suffering from dermatologic condition in the treatment area or has a significant scar in the hair treatment area that, in the opinion of the investigator, will make hair growth difficult (such as systemic burns, etc.).
6. History of autoimmune disease or organ transplantation or a patient on immunosuppressive medication(s).
7. Diagnosis of cancer, receiving active treatment
8. Active systemic infection
9. Requires chronic antibiotics, systemic corticosteroids
10. Use of systemic agents that increase bleeding or clotting, or disorders associated with these effects, including patients receiving GIIB/IIIa inhibitors within 2 weeks prior to the study procedure through to 1 week after the study procedure.
11. Clinically significant medical or psychiatric illness currently or within 30 days of study screening as determined by the investigator
12. Prior surgery in the treatment area
13. Any disease or condition (medical or surgical) that, in the opinion of the investigator, might compromise dermatologic, hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system function; or any condition that would place the subject at increased risk
14. Pregnant or lactating women or women trying to become pregnant
15. Known allergic reaction to components of study treatment and/or study injection procedure
16. Subject has any disorder that may prevent compliance to study procedures and visits
17. Subject who is part of the study staff, a family member or friend
18. Diabetes or thyroid disorder
19. Subject who has a sensitive, irritated, or abraded scalp area.
20. Women who have an alternate diagnosis that is associated with hair loss.
21. Body Mass Index < 18kg/m2
22. Clinically significant abnormal findings on laboratory screening panels, including hemoglobin ≤ 10 g/dL.
23. Hepatic dysfunction, as defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin levels > 1.5 times the upper limit of normal range (x ULN) prior to randomization.
24. Chronic renal insufficiency as defined as a serum creatinine > 1.2 mg/dL for women and > 1.5 mg/dL for men.
25. An elevated PT/PTT, INR, or platelet count < 100 x 109/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ken Washenik, MD, Principal Investigator — Bosley Medical/NYU
Locations (4):
- United States (4):
  - Tower Outpatient Surgery Center--Dr. Joel Aronowitz, Los Angeles, California
  - Foundation For Hair Restoration, Miami, Florida
  - Glasgold Surgery Group, Highland Park, New Jersey
  - Laser & Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Festa E, Fretz J, Berry R, Schmidt B, Rodeheffer M, Horowitz M, Horsley V. Adipocyte lineage cells contribute to the skin stem cell niche to drive hair cycling. Cell. 2011 Sep 2;146(5):761-71. doi: 10.1016/j.cell.2011.07.019. PMID 21884937
- [Background] Zhu M, Zhou Z, Chen Y, Schreiber R, Ransom JT, Fraser JK, Hedrick MH, Pinkernell K, Kuo HC. Supplementation of fat grafts with adipose-derived regenerative cells improves long-term graft retention. Ann Plast Surg. 2010 Feb;64(2):222-8. doi: 10.1097/SAP.0b013e31819ae05c. PMID 20098110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control
Started | 16 | 22 | 24 | 9
Completed | 12 | 19 | 21 | 8
Not Completed | 4 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All subjects were included in the analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control | Total
Number analyzed (Participants) | 16 | 22 | 24 | 9 | 71
Age, Customized [Mean (Standard Deviation); unit: years]
  Age(Years) | 40.0 (9.1) | 43.1 (13.3) | 40.5 (12.7) | 36.1 (5.4) | 40.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7 | 3 | 17
  Male | 14 | 17 | 17 | 6 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12 | 4 | 28
  Not Hispanic or Latino | 8 | 16 | 12 | 5 | 41
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 3
  White | 15 | 21 | 22 | 9 | 67
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety & Tolerability Assessment of SAE/AE
Description: Safety & Tolerability of Experimental Treatment (ADRC) Assessment of SAE/AE
Time Frame: Enrollment to 52 weeks
Measure: Number; unit: events
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control
Number analyzed (Participants) | 16 | 22 | 24 | 9
events
  Total Number of Adverse Events | 5 | 9 | 12 | 2
  Unanticipated Adverse Eventss | 0 | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0 | 0

2. Secondary Outcome: Terminal (Non-Vellus) Hair Count--Change From Baseline
Description: Terminal (Non-Vellus) Hair Count Assessment by Macrophotography
Time Frame: Enrollment to 52 weeks
Population: mITT, Baseline Norwood-Hamilton III
Measure: Mean (Standard Error); unit: Hairs
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control
Number analyzed (Participants) | 6 | 11 | 5 | 4
Hairs | -5.62 (6.09) | 16.2 (4.98) | -0.57 (7.53) | -7.92 (8.98)
Statistical Analysis 1: Comparison: Fat + Low Dose ADRC vs No Fat Control; Test type: Superiority; p = 0.032, ANCOVA
Statistical Analysis 2: Comparison: Fat + Low Dose ADRC vs No Fat Control; Non-vellus hair count in the low-dose ADRC group in the NW3 subgroup beginning at Week 6 (mean change from baseline persisting through weeks 12 , 24, and 52; Test type: Other; p = 0.0318, ANCOVA — P value cited is the difference in non-vellus hair count between the low-dose ADRC NW3 group and the no-fat saline control at week 24

3. Secondary Outcome: Hair Satisfaction Questionnaire Responses at Week 24 for Questions 1 Through 4
Description: Percent of positive responses, defined by increase of 1 or more from baseline, on specific written assessment of treatment outcome by Investigators scored 1-5, value 1 is lowest, value of 5 is highest, higher values represent more positive responses
Time Frame: Enrollment to 24 weeks
Population: The Baseline NW3 subgroup included all male subjects with baseline Norwood Scale III, III-A and III-V.
Measure: Number; unit: % of participants with + responses
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control
Number analyzed (Participants) | 6 | 7 | 12 | 3
% of participants with + responses | 12.5 | 34.4 | 20.8 | 4.1

ADVERSE EVENTS:
Time Frame: From Enrollment through 52 Weeks
Description: Events were reported by Investigators, which was supplemented by information from study subjects to Investigators. Attribution was performed by study Medical Director. No adverse Events were attributed to the experimental procedure / product.
Arm/Group | Fat + High Dose ADRC | Fat + Low Dose ADRC | Fat Alone | No Fat Control
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/22 | 0/24 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/22 | 0/24 | 0/9
Other Adverse Events (participants affected / at risk) | 5/16 | 9/22 | 11/24 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat + High Dose ADRC (N=16) | Fat + Low Dose ADRC (N=22) | Fat Alone (N=24) | No Fat Control (N=9)
Brusing or Edema (Skin and subcutaneous tissue disorders) | 5 (5) | 8 (8) | 11 (11) | 2 (2) — At liposuction or donor site, with or without pain
Shilgles (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hickups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT02503852/Prot_SAP_000.pdf